CLINICAL TRIAL: NCT00617162
Title: A Clinical Evaluation for the Management of Patients With Major Depressive Disorder, Single or Recurrent Episode, With Deep Brain Stimulation
Brief Title: Deep Brain Stimulation for Major Depressive Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business reasons
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-07-01
Record Dates: First submitted 2007-12-26; First posted 2008-02-15 (Estimated); Results first posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Depressive Disorder, Major; Unipolar Depression
Keywords: C-07-01, BROADEN™, Deep Brain Stimulation, Major Depressive Disorder, Unipolar Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DBS Active Treatment Group (Experimental): Deep Brain Stimulation, Libra Deep Brain Stimulation System: DBS Active Treatment Group - implanted with investigational device and activated for stimulation
  Interventions: Device: Deep Brain Stimulation, Libra Deep Brain Stimulation System
- DBS Control Group (Placebo Comparator): Deep Brain Stimulation, Libra Deep Brain Stimulation System: implanted with investigational device, but will not receive active stimulation for the first 6 months of the study
  Interventions: Device: Deep Brain Stimulation, Libra Deep Brain Stimulation System

INTERVENTIONS:
Device: Deep Brain Stimulation, Libra Deep Brain Stimulation System — DBS Active Treatment Group - implanted with investigational device and activated for stimulation
  Other Names: Libra Deep Brain Stimulation System
  Arms: DBS Active Treatment Group
Device: Deep Brain Stimulation, Libra Deep Brain Stimulation System — implanted with investigational device, but will not receive active stimulation for the first 6 months of the study
  Other Names: Libra Deep brain Stimulation System
  Arms: DBS Control Group

SUMMARY:
This study is designed as a prospective, multi-centered, double-blind, randomized, controlled 12-month pivotal study to evaluate the safety and efficacy of the ANS Libra® Deep Brain Stimulation System for patients with major depressive disorder who have failed at least 4 treatments in the current episode. The primary outcome assessment will occur at 6 months: however, all patients will be followed for 1 year. A total of 201 patients will be randomized from up to 20 sites.

Each potential patient will be pre-screened according to the inclusion/exclusion criteria. A narrative of what study participation entails, will be used to educate potential participants on study requirements. Prior to on-site baseline evaluations, the patient will sign the informed consent. Patients will then undergo 3 baseline evaluations, with each of these evaluations to occur no less than 2 weeks apart from each other. The first 2 baseline visit evaluations will be performed by separate psychiatrists in order to confirm the patient's diagnosis. All patients will be scheduled for surgery, to occur no less than two weeks and no more than 1 month after final baseline evaluation, to implant the ANS Libra® Deep Brain Stimulation system. After device implantation, patients will be randomly assigned to 1 of 2 groups in a 2:1 ratio (Active Treatment Group & Control Group).

After system implant (Week 0), the patient will return to clinic approximately 2 weeks after surgery for evaluation and treatment randomization into either Group 1 or Group 2 (Group 1 = Active Treatment Group; Group 2 = Control Group). Patient will then return to clinic for subsequent evaluations at 2 weeks, 4 weeks, 6 weeks, 8 weeks, 3 months, 4 months, 5 months, 6 months, 7 months, 8 months, 9 months, 10 months, 11 months, and 1 year post system implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women (non-pregnant) age is 21-70 years;
2. Diagnosed with non-psychotic major depressive disorder, single or recurrent episode by DSM-IV-TR criteria derived from the MINI;
3. First episode onset before age 45;
4. Current episode ≥ 12 months duration;
5. In the current episode: Documented resistance (i.e.persistence of the major depressive episode) to a minimum of 4 adequate depression treatments from at least 3 different treatment categories (e.g. SSRI's, SNRI's, TCA's, MAO inhibitors, Mirtazipine, Nefazodone, Trazodone, Bupropion, lithium augmentation, thyroid augmentation, ECT); Adequacy of treatments as defined by a score of at least 3 according to the amended Antidepressant Treatment History Form (ATHF) criteria;
6. In Lifetime: Received a course of psychotherapy for depression;
7. Montgomery Asberg Depression Rating Scale (MADRS) of ≥ 22 at 3 separate baseline visits, rated by 2 separate psychiatrists, Baseline 2 and Baseline 3 MADRS scores cannot be separated by > 6 weeks and cannot improve ≥ 20%;
8. Global Assessment of Function, score <50;
9. Modified mini-mental state examination (MMSE) score ≥24;
10. No change in current antidepressant medication regimen or medication free ≥4 weeks prior to study entry (with exception to sleep, cholesterol, blood pressure, sexual dysfunction, non-migraine headache medication, or medication for other medical reasons not related to depression, in which changes to dose or type will be allowed during course of study);
11. Able to give informed consent in accordance with institutional policies;
12. Able to comply with all testing and follow-up requirements as defined by the study protocol;
13. Must be determined medically stable by surgeon, to undergo deep brain stimulation surgical procedure.
14. Must have platelet count, PT and PTT within normal limits of the laboratory.
15. During last 6 months in the current episode documented treatment under the care of a licensed psychiatrist/psychologist.

Exclusion Criteria:

1. A diagnosis of a bipolar I or bipolar II disorder by DSM-IV-TR criteria, derived from the MINI;
2. Meets criteria for borderline or antisocial personality disorder in the last 12 months by DSM-IV-TR criteria, derived from the Cluster B Personality Disorders Sections 301.7 - 301.83, and screened via SCID-II at Baseline visit;
3. In the current depressive episode, has been diagnosed with General Anxiety Disorder (GAD) - as defined by the DSM-IV-TR, and GAD is the primary diagnosis;
4. Has an intracranial Central Nervous System (CNS) disease that impairs motor, sensory or cognitive function or that requires intermittent or chronic medication (e.g., Parkinson's Disease, chronic migraine, stroke, Huntington's, head trauma, etc.) with exception to non-migraine headaches;
5. Has been diagnosed with fibromyalgia or has a current condition which requires chronic pain narcotic usage (e.g. morphine, methadone);
6. Has been currently diagnosed with chronic fatigue syndrome;
7. Substantial suicidal risk as defined by (1) MADRS item 10 score of 5 or 6, (2) a current plan and intent,(3) clinician judgment that there is a clear immediate intent for self-harm, (4) more than 3 suicide attempts within the last 12 months;
8. Co-morbid obsessive compulsive disorder, posttraumatic stress disorder, panic disorder, bulimia or anorexia nervosa if previously present, must be in remission for 6 months as defined by DSM-IV-TR criteria, derived from the MINI;
9. Alcohol, medication, or illegal substance dependence or abuse within last 12 months derived from the MINI;
10. Diagnosis of sleep apnea confirmed by a sleep test that is not adequately treated;
11. Advanced cardiovascular disease which renders anesthesia and surgery as unsafe as determined by neurosurgeon;
12. Clinically relevant abnormality (e.g. tumor or growth) on study MRI;
13. Has cardiac pacemaker/defibrillator or other implanted active stimulator;
14. Has a medical condition requiring a repetitive MRI body scan;
15. Requires chemotherapy for the treatment of malignancy or requiring chronic oral or intravenous (immunosuppressive or) steroid therapy;
16. Is unable to comply with study visit schedule and timeline;
17. Past ablative or relevant intracranial surgery;
18. A female lactating or of child bearing potential, with a positive pregnancy test or not using adequate contraception;
19. Lifetime psychotic disorders, schizophrenia, or schizoaffective disorder defined by DSM-IV-TR;
20. Psychotic features in current depressive episode as diagnosed by DSM-IV-TR criteria;
21. Other medical conditions likely to require hospitalization within the next year;
22. Received ECT within 3 months prior to enrollment, or requires ECT for the duration of the study;
23. Has a history of epilepsy or history of status epilepticus;
24. Plans to use diathermy;
25. Has any metallic implants such as aneurysm clips or cochlear implants;
26. Currently participating in another investigational device, drug or surgical trial

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2008-03; Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: DeLea Peichel, Study Director — Abbott Medical Devices
Locations (13):
- United States (11):
  - Stanford University School of Medicine, Stanford, California
  - Alexian Brothers Behavioral Health Hospital, Chicago, Illinois
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - The Zucker Hillside Hospital, Glen Oaks, New York
  - Columbia University Medical Center, New York, New York
  - Medical Univeristy of South Carolina (MUSC), Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Neuroscience Institute, Seattle, Washington
- University of British Columbia, Vancouver, British Columbia, Canada
- University of Dundee, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holtzheimer PE, Husain MM, Lisanby SH, Taylor SF, Whitworth LA, McClintock S, Slavin KV, Berman J, McKhann GM, Patil PG, Rittberg BR, Abosch A, Pandurangi AK, Holloway KL, Lam RW, Honey CR, Neimat JS, Henderson JM, DeBattista C, Rothschild AJ, Pilitsis JG, Espinoza RT, Petrides G, Mogilner AY, Matthews K, Peichel D, Gross RE, Hamani C, Lozano AM, Mayberg HS. Subcallosal cingulate deep brain stimulation for treatment-resistant depression: a multisite, randomised, sham-controlled trial. Lancet Psychiatry. 2017 Nov;4(11):839-849. doi: 10.1016/S2215-0366(17)30371-1. Epub 2017 Oct 4. PMID 28988904

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The aim of this prospective, multi-centered, double-blind, randomized, controlled 12-month pivotal study is to evaluate the safety and efficacy of the SJM Libra® Deep Brain Stimulation System for patients with major depressive disorder who had failed at least 4 treatments in the current episode. The primary outcome assessment occurred at the 6 month vistit, however all patients were followed for 1 year. A total of 201 patients were to be randomized from up to 20 sites.
Pre-assignment Details: The protocol allowed enrollment during the screening period. 125 were enrolled but only 90 continued on to receive DBS implants.
Period: Overall Study
Arm/Group | DBS Active Treatment Group | DBS Control Group
Started | 60 | 30
Completed | 53 | 27
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DBS Active Treatment Group | DBS Control Group | Total
Number analyzed (Participants) | 60 | 30 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.53 (9.73) | 48.70 (10.56) | 49.62 (10.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 17 | 47
  Male | 30 | 13 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 58 | 26 | 84
  African American | 0 | 1 | 1
  Hispanic | 2 | 3 | 5
  Asian | 0 | 0 | 0
  Other | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 2 | 6
  United States | 55 | 27 | 82
  United Kingdom | 1 | 1 | 2
Montgomery and Asberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: units on a scale] — The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60.
  units on a scale | 33.8 (4.48) | 37.3 (3.82) | 35.5 (4.15)

OUTCOME MEASURES:

1. Primary Outcome: Montgomery and Asberg Depression Rating Scale (MADRS) Score at Baseline and the Average of Months 4, 5, and 6
Description: The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60. The lower a score the less symptom severity is seen.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBS Active Treatment Group | DBS Control Group
Number analyzed (Participants) | 60 | 30
score on a scale
  Mean Baseline | 33.8 (4.48) | 37.3 (3.82)
  Mean of Months 4, 5, 6 | 27.5 (9.73) | 29.4 (9.52)
Statistical Analysis 1: Comparison: DBS Active Treatment Group vs DBS Control Group; Test type: Superiority; p = 0.3989, Fisher Exact; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-5.5 to 2.2]

2. Secondary Outcome: Baseline MADRS to MADRS at 1 Year
Description: as for outcome 1
Time Frame: Baseline to 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBS Active Treatment Group | DBS Control Group
Number analyzed (Participants) | 60 | 30
score on a scale
  Baseline MADRS | 33.8 (4.48) | 37.3 (3.82)
  Mean MADRS at 12 months | 23.2 (12.15) | 26.7 (12.06)

3. Secondary Outcome: Number of Participants With Adverse Events (i.e., Hospitalization Due to Worsening Depression, Suicidal Ideation or Behavior, Medical Treatment, and Device Related Events) That Occur Over Study Duration
Time Frame: 6 months-1 year
Measure: Count of Participants; unit: Participants
Arm/Group | DBS Active Treatment Group | DBS Control Group
Number analyzed (Participants) | 60 | 30
Participants
  0 adverse events | 35 | 12
  1 adverse event | 13 | 12
  2 adverse events | 6 | 2
  3 adverse events | 3 | 1
  4 adverse events | 1 | 2
  5 adverse events | 2 | 0
  7 adverse events | 0 | 1

4. Secondary Outcome: Global Assessment Scale (GAF) Score at Baseline and 1 Year
Description: The Global Assessment Scale (GAF) is a hypothetical continuum of mental health illness that looks at psychological, social, and occupational functioning. It measures how much a person's symptoms affect their day to-day life on a scale of 0 to 100. A score of 100-91 indicates no symptoms, 90-81 indicates absent minimal symptoms, 80-71 indicates symptoms that are transient and reactions expectable to psychosocial stressors, 70-61 indicates mild symptoms, 60-51 indicates moderate symptoms, 50-41 indicates serious symptoms, 40-31 indicates some impairment in reality testing or communication OR major impairment in several areas, 30-21 indicates delusions or hallucinations, 20-11 indicates danger of hurting self or others OR occasionally fails to maintain personal hygiene, 10-1 indicates persistent danger of severely hurting self or others OR persistent inability to maintain minimal personal hygiene OR serious suicidal act with clear expectation of death and 0 indicates inadequate data.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBS Active Treatment Group | DBS Control Group
Number analyzed (Participants) | 60 | 30
score on a scale
  Baseline GAF | 42.0 (4.27) | 40.6 (4.73)
  Month 12 GAF | 54.2 (15.99) | 53.7 (13.34)

5. Secondary Outcome: Hamilton Rating Scale for Depression - 17 Item (HRSD-17) Score at Baseline and 6 Months
Description: The Hamilton Rating Scale for Depression - 17 item (HDRS-17) ranging from 0-52 used to assess potential changes in the severity of depressive symptoms (Hamilton 1960; Hamilton 1967). It is used to evaluate depressed mood, vegetative and cognitive symptoms of depression, and co-morbid anxiety symptoms. Scoring is based on the 17-itemscale and scores of 0-7 are considered as being normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression; the maximum score being 52 on the17-point scale.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DBS Active Treatment Group | DBS Control Group
Number analyzed (Participants) | 56 | 29
units on a scale
  Baseline HDRS-17 | 20.3 (3.78) | 22.6 (4.44)
  HDRS-17 Month 6 | 17.5 (7.57) | 19.0 (7.94)

6. Secondary Outcome: Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) Score From Baseline to 1 Year
Description: The Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) is a self-report instrument designed to measure the degree of enjoyment and satisfaction experienced by subjects in various areas of daily functioning. There are 16 areas of functioning, each scored from 1 (very poor) to 5 (very good). The range of scores is 16-80, with lower scores representing lower functioning and satisfaction.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBS Active Treatment Group | DBS Control Group
Number analyzed (Participants) | 58 | 28
score on a scale
  Baseline Q-LES-Q | 33.5 (6.08) | 28.5 (5.87)
  12 Month Score Q-LES-Q | 40.1 (10.72) | 36.8 (11.35)

7. Secondary Outcome: Inventory of Depressive Symptomology (IDS-C30) Score From Baseline to 1 Year
Description: The construction of the Inventory of Depressive Symptomology (IDS-C30) was intended to remedy deficits in the Hamilton Scale for Depression (HRSD-17) and Montgomery and Asberg (MADRS) depression rating scales by, among others, including all nine symptom domains needed to diagnose a DSM-IV major depressive episode in order to assess symptom remission, improve ability to detect milder levels of symptoms than the HRSD-17, and provide unconfined and more equivalent weighting among items. There are two versions of the IDS with identical items: a clinician rating (IDS-C30) and a self-report (IDS-SR30). Each of the 30 items is rated from 0 to 3, with increasing severity represented by a higher rating. (Rush et al. 1996). When complete, the IDS-C30 and IDS-SR30 are scored by summing responses to 28 of the 30 items to obtain a total score ranging from 0 to 84. Either appetite increase or decrease, but not both, are used to calculate the total score.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBS Active Treatment Group | DBS Control Group
Number analyzed (Participants) | 60 | 30
score on a scale
  Baseline IDS | 37.0 (7.42) | 41.1 (38.24)
  Month 12 IDS | 26.5 (13.87) | 31.2 (14.29)

8. Secondary Outcome: Quick Inventory of Depressive Symptomatology (QIDS-SR) Scores From Baseline to 1 Year
Description: The Quick Inventory of Depressive Symptomatology Self Report (QIDS- SR) is a 16-question shortened self-test, derived from the 30-item IDS. Questions in the QIDS - SR-116 correlate with the nine DSM-IV symptom criterion domains, including: Sleep disturbance (initial, middle, and late insomnia or hypersomnia) (Q 1 - 4), Sad mood (Q 5), Decrease/increase in appetite/weight (Q 6 - 9), Concentration (Q 10), Self-criticism (Q 11), Suicidal ideation (Q 12), Interest (Q 13), Energy/fatigue (Q 14), Psychomotor agitation/retardation (Q 15 - 16). The severity of depression can be judged based on the total score ranging from 1-27. A score of 1-5 indicates No depression, 6-10 indicates Mild depression,11-15 indicates Moderate depression, 16-20 indicates Severe depression and 21-27 indicates Very severe depression.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBS Active Treatment Group | DBS Control Group
Number analyzed (Participants) | 60 | 30
score on a scale
  Baseline QIDS-SR | 17.4 (3.28) | 19.5 (2.70)
  Month 12 QIDS-SR | 12.8 (6.91) | 14.1 (6.01)

9. Secondary Outcome: Work and Social Adjustment Scale (WSAS) Score From Baseline to 1 Year
Description: The WSAS is a modification of a scale introduced by Hafner and Marks (1976), consisting of 0-8 point ratings of the extent to which symptoms interfere with five areas of daily functioning: work, home management, private leisure, social leisure, and family relationships. It is a well-validated, widely used self-report measure. Additional time points include weeks 4, 8, 12, 16, and 40. A total score calculated as a sum of all items (possible range 0-40) was used in the analyses with higher scores indicating more impairment.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBS Active Treatment Group | DBS Control Group
Number analyzed (Participants) | 60 | 30
score on a scale
  Baseline WSAS | 32.9 (4.66) | 35.2 (3.06)
  12 month WSAS | 25.5 (11.46) | 29.6 (9.45)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | DBS Active Treatment Group | DBS Control Group
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/30
Serious Adverse Events (participants affected / at risk) | 23/60 | 7/30
Other Adverse Events (participants affected / at risk) | 40/60 | 24/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DBS Active Treatment Group (N=60) | DBS Control Group (N=30)
Bariatric weight loss surgery (Surgical and medical procedures) | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 2 | 0
Elective admission to IP unit to alleviate burden on primary carer (General disorders) | 1 | 0
Patient re-admitted on an elective basis to IP unit (General disorders) | 1 | 0
Infection (Infections and infestations) | 5 | 1
Post-operative discomfort (Surgical and medical procedures) | 1 | 0
Seizure or convulsion (General disorders) | 1 | 1
Suicide or suicide attempt (Psychiatric disorders) | 2 | 2
Increase in depressive symptoms (Psychiatric disorders) | 10 | 2
Hearing and visual disturbance (General disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 0
General erosion (Infections and infestations) | 1 | 0
Headache (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DBS Active Treatment Group (N=60) | DBS Control Group (N=30)
Headache (General disorders) | 18 | 10
Middle back pain (General disorders) | 0 | 1
Generalized body pain (General disorders) | 0 | 1
Hyperphagia (General disorders) | 0 | 1
Feeling hot constant (General disorders) | 1 | 0
Feeling cold constant (General disorders) | 1 | 0
Mild worsening of pre-existing tremor (General disorders) | 1 | 0
Jaw pain (General disorders) | 1 | 0
Cutting self (General disorders) | 0 | 1
Suicidal ideation (General disorders) | 0 | 1
Peripheral neuropathy (General disorders) | 1 | 0
Nocturia with urinary frequency (General disorders) | 1 | 0
Dyspepsia (General disorders) | 1 | 0
Flu syndrome (General disorders) | 1 | 0
Leg cramps and soreness on legs (General disorders) | 1 | 0
Motor incoordination left side (General disorders) | 1 | 0
Fractured arm (General disorders) | 0 | 1
Feeling of surgical pressure on IPG site (General disorders) | 0 | 1
Mild tremor (General disorders) | 1 | 0
Oral Thrush (General disorders) | 1 | 0
Churning feeling in the head (General disorders) | 0 | 1
Irritability (General disorders) | 1 | 0
Ridge right side of scalp with twinges of pain (General disorders) | 1 | 0
Burned self left deltoid area (General disorders) | 1 | 0
Increased irritability (General disorders) | 0 | 1
Chest pressure (General disorders) | 0 | 1
Occasional, very mild tremor (General disorders) | 0 | 1
Back pain from carrying heavy load of water (General disorders) | 1 | 0
Patient claims she can "feel the wires in brain" (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Unilateral eye swelling (General disorders) | 0 | 1
Pustule on suture line (General disorders) | 0 | 1
Hypercholesterolaemia (General disorders) | 1 | 0
Reports of increased cravings for chocolate and biscuits (General disorders) | 1 | 0
Complaining of aches and pains and cramps in hands, arms, and feet (General disorders) | 1 | 0
Infection (Infections and infestations) | 2 | 3
Post operative discomfort (General disorders) | 5 | 2
Cerebrospinal fluid leakage (General disorders) | 0 | 1
Post-operative pain (General disorders) | 6 | 6
Subcutaneous hemorrhage or seroma (General disorders) | 1 | 2
Aphasia (General disorders) | 1 | 0
Nausea and/or vomiting (General disorders) | 4 | 4
Sleep disturbance (General disorders) | 4 | 6
Pulling sensation along extension site (General disorders) | 6 | 1
Persistent pain or redness at the IPG site or surgery site/extension (General disorders) | 1 | 7
Cerebrospinal fluid abnormality (General disorders) | 0 | 1
Hearing and visual disturbance (General disorders) | 9 | 0
Disequilibrium (General disorders) | 4 | 1
Increase in depressive symptoms (General disorders) | 4 | 4
Anxiety (General disorders) | 6 | 7
Eye disorder (General disorders) | 2 | 2
Neuralgia (General disorders) | 5 | 0
Drowsiness (General disorders) | 3 | 0
Skin disorder (General disorders) | 2 | 3
General erosion or local skin erosion over the IPG, burr hold cap, and/or extension (General disorders) | 9 | 1
Paresthesia (General disorders) | 2 | 6
Hypomania (Psychiatric disorders) | 0 | 2
Pneumonia (General disorders) | 0 | 1
Suicide or suicide attempt (Psychiatric disorders) | 0 | 1
Sweating (General disorders) | 2 | 0
Diarrhea (General disorders) | 2 | 2
Cognitive impairment (General disorders) | 2 | 1
Rapid heart rate (General disorders) | 0 | 2
Increase in drug side effects (General disorders) | 2 | 2
Myoclonus (General disorders) | 1 | 0
Syncope (General disorders) | 0 | 1
Asthenia, hemiplegia, or hemiparesis (General disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Attention deficit (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/62/NCT00617162/Prot_SAP_000.pdf